CLINICAL TRIAL: NCT01295905
Title: Prospective Study of an Investigational Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-347-C-004
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- delefilcon A (Experimental): Investigational contact lenses worn in both eyes on a daily wear, daily disposable basis for 3 months.
  Interventions: Device: delefilcon A contact lens
- narafilcon B (Active Comparator): Commercially marketed contact lenses worn in both eyes on a daily wear, daily disposable basis for 3 months.
  Interventions: Device: narafilcon B contact lens

INTERVENTIONS:
Device: delefilcon A contact lens — Investigational silicone hydrogel, single vision soft contact lens
  Arms: delefilcon A
Device: narafilcon B contact lens — Commercially marketed silicone hydrogel, single vision soft contact lens
  Arms: narafilcon B

SUMMARY:
The purpose of this study is to evaluate the performance of an investigational daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal eyes who are not using any ocular medications.
* Be of legal age of consent and sign Informed Consent document. If under legal age of consent, legally authorized representative must sign Informed Consent document and subject must sign Assent document.
* Willing and able to wear spherical contact lenses for at least 5 days per week.
* Willing and able to wear spherical contact lenses within the available range of powers of -1.00 diopter(D) to -6.00D in 0.25D steps.
* Best spectacle-corrected visual acuity greater than or equal to 20/25.
* Manifest cylinder less than or equal to 0.75D.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any active anterior segment ocular disease that would contraindicate contact lens wear.
* Any use of systemic medications for which contact lens wear could be contraindicated as determined by the investigator.
* History of refractive surgery or irregular cornea.
* History of pathologically dry eye.
* Eye injury within twelve weeks immediately prior to enrollment for this trial.
* Currently enrolled in any clinical trial.
* Participation in a contact lens or contact lens care product clinical trial within the previous 30 days.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from six (6) US study centers.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | Delefilcon A | Narafilcon B
Started | 60 | 30
Completed | 58 | 30
Not Completed | 2 | 0
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — Met exclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delefilcon A | Narafilcon B | Total
Number analyzed (Participants) | 60 | 30 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 29.01 (8.86) | 31.39 (10.05) | 29.80 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 19 | 59
  Male | 20 | 11 | 31
Region of Enrollment [Number; unit: participants]
  United States | 60 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Corrected Distance Monocular Visual Measurement in Normal Illumination Reported as Visual Acuity
Description: Each eye tested individually while reading a chart distant to the participant in normal lighting. Visual acuity was measured using a Snellen chart, with 20/20 Snellen acuity considered normal distance-eyesight. Visual acuity is reported as the number of eyes achieving 20/20 Snellen acuity or better.
Time Frame: 3 months of wear, lenses replaced daily
Population: Per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 58 | 30
Number analyzed (eyes) | 116 | 60
eyes | 111 | 58

2. Secondary Outcome: Overall Vision
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 3 months of wear time. Overall vision was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 3 months of wear, lenses replaced daily
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 58 | 30
Units on a scale | 9.5 (0.8) | 9.1 (1.1)

3. Secondary Outcome: Overall Comfort
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 3 months of wear time. Overall comfort was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 3 months of wear, lenses replaced daily
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 58 | 30
Units on a scale | 9.3 (0.9) | 8.9 (1.2)

4. Secondary Outcome: Overall Handling
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 3 months of wear time. Overall handling was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 3 months of wear, lenses replaced daily
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 58 | 30
Units on a scale | 9.1 (1.3) | 9.1 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 19-JAN-2011 to 20-MAY-2011.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Delefilcon A | Narafilcon B
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/30
Other Adverse Events (participants affected / at risk) | 0/60 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delefilcon A (N=60) | Narafilcon B (N=30)
Sterile infiltrate with secondary iritis (Eye disorders) | 0 | 1 — One eye. Resolved. Resumed wearing study lenses and completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.